CLINICAL TRIAL: NCT00589732
Title: Valsartan for SUPpression of Plaque Volume and Restenosis After Drug-Eluting Stent (The VAL-SUPPRESS TRial)
Brief Title: Valsartan for Suppression of Plaque Volume and Restenosis After Drug-Eluting Stent
Acronym: VAL-SUPPRES
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seung-Jung Park (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, M.D., Ph.D.,Professor of Medicine Asan Medical Center, University of Ulsan, College of Medicine, CardioVascular Research Foundation, Korea
Organization: CardioVascular Research Foundation, Korea (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0077
Record Dates: First submitted 2007-12-31; First posted 2008-01-10 (Estimated); Last update posted 2012-08-08 (Estimated); Status verified 2012-08

CONDITIONS: Coronary Artery Disease
Keywords: stents; angiotensin-converting enzyme
MeSH Terms: conditions — Coronary Artery Disease | interventions — Valsartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Valsartan treatment gorup (Experimental): Valsartan 160mg per day group
  Interventions: Drug: Valsartan
- No Valsartan treatment group (No Intervention): No valsartan treatment

INTERVENTIONS:
Drug: Valsartan — Valsartan 160mg per day
  Arms: Valsartan treatment gorup

SUMMARY:
To evaluate that angiotensin-converting enzyme (ACE) inhibitors and angiotensin-converting enzyme receptor blockers (ARBs) reduce the risk of restenosis after DES implantation.

DETAILED DESCRIPTION:
Stimulation of the angiotensin II type 1 (AT1) receptors after arterial injury promotes vascular smooth muscle cell (VSMC) migration, proliferation, and extracellular matrix production, leading to the hope that blockade of this receptor by angiotensin-converting enzyme inhibitors (ACEI) or specific (AT1) receptor antagonists (ARBs) might reduce intimal hyperplasia. However, despite confirmatory evidence in several animal models of restenosis, the large scale MERCATOR and MARCATOR trials of cilazapril with balloon angioplasty failed to show benefit. In 1999, Kondo reported the results of a randomized pilot trial of 100 patients who received Palmaz-Schatz stents and were randomized to receive the ACE inhibitor quinapril or placebo. The volume of neointimal hyperplasia assessed by IVUS was significantly less quinapril than the control group (18 ± 0.6 mm3 vs. 25 ± 0.6 mm3; p < 0.05). The quinapril group's restenosis rate was 16%, with the quinapril benefit being observed only in patients with the D/D and I/D genotypes. Also, other study reported on a consecutively treated cohort of 1,598 stented patients, noting that ACE inhibitor usage at the time and after stenting reduced the risk of subsequent revascularization dramatically (adjusted odds ratio, 0.46; p = 0.001). In the ValPREST trial which is a single-center randomized trial of patients receiving stents for type B2/C lesions, comparing valsartan (and ARV) 80 mgs daily with open treatment, patients randomized to valsartan had a 19% incidence of restenosis compared with 39% in the open treatment arm (p = 0.005).

Recently, several randomized studies were conducted to compare the safety and efficacy of the two leading drug-eluting stent (DES). However, data on the association of ARBs for suppression of neointimal hyperplasia are limited in the DES era. Therefore, a pivotal randomized study is warranted.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical 1) Patients with angina and documented ischemia or patients with documented silent ischemia 2) Patients who are eligible for intracoronary stenting 3) Age >18 years, <75 ages 4) Preserved left ventricular ejection fraction (>40%) 5) Written informed consent to the study protocol 6) Patients with hemodynamic stability and appropriate blood pressure, which were suitable for administration of valsartan 160mg
2. Angiographic: Patients who have

1) Significant ischemic narrowing (target vessel)

1. De novo coronary lesion (no restriction of lesion length)
2. Percent diameter stenosis ≥50% by visual estimate
3. Reference vessel size ≥2.5 mm by visual estimation
4. Lesions suitable for stenting

And/Or

2) Non-significant non-ischemic intermediate narrowing (non-target vessel)

1. Percent diameter stenosis 20%~50% by visual estimate
2. No objective evidence of ischemia

Exclusion Criteria:

1. Patients received a Angiotensin converting enzyme inhibitor (ACE-I) or ACE-receptor blockers (ARBs) in the previous week prior to enrollment
2. History of bleeding diathesis or coagulopathy
3. Pregnant
4. Known hypersensitivity or contra-indication to contrast agent and heparin
5. Limited life-expectancy (less than 1 year)
6. Acute ST-elevation myocardial within 1 week
7. Characteristics of lesion 1) Left main disease 2) In-stent restenosis 3) Graft vessels
8. Hematological disease (Neutropenia <3000/mm3, Thrombocytopenia <100,000/mm3)
9. Hepatic dysfunction, liver enzyme (ALT and AST) elevation >3 times normal
10. Renal dysfunction, creatinine >2.0mg/dL
11. Contraindication to aspirin and clopidogrel

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2006-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Angiographic in-stent late-loss (target vessel) | at 8-month follow-up.

SECONDARY OUTCOMES:
Composite of Major cardiac adverse events including death, Q-MI, Non Q-MI, and target lesion or vessel revascularization -Delta change in percent atheroma area and volume | 30 days
Composite of Major cardiac adverse events including death, Q-MI, Non Q-MI, and target lesion or vessel revascularization | 9 months
Each component of MACE | 3 days in average
  3 day hospitalization is normal for index procedure and outcome needs to be measured at discharge.
Each component of MACE | 30 days
Each component of MACE | 9 months
In-stent and in-segment restenosis rate | 8 months
In-segment late loss | 8 months
Percent atheroma volume of 10mm length by IVUS examination (non-target vessel) in IVUS-substudy | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Jung Park, MD, PhD, Principal Investigator — Department of Medicine, Asan Medical Center, University of Ulsan College of Medicine
Locations (5):
- South Korea (5):
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - St. Mary's Catholic Medical Center, Seoul
  - Yonsei University Medical Center, Seoul
  - Ajou University Hospital, Suwon